CLINICAL TRIAL: NCT06024200
Title: Effect of Whole-process Transcutaneous Electrical Acupoint Stimulation on Opioid Consumption After Gastrointestinal Laparoscopic Surgery: a Prospective, Randomised, Blinded, Placebo-controlled Study
Brief Title: Transcutaneous Electrical Acupoint Stimulation for Opioid Consumption After Gastrointestinal Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFEC-2023-327
Record Dates: First submitted 2023-08-16; First posted 2023-09-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Transcutaneous Electrical Acupoint Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole-process transcutaneous electrical acupoint stimulation (Experimental): Electrical stimulation is performed within 24h before surgery, 30min before anesthesia induction and 3 days after surgery, each stimulation was 30min. Patients are treated bilaterally at two groups of distal acupoints: one group consisted of Hegu (LI4) and Neiguan (PC6), the other contained Zusanli (ST36) and Shanyinjiao (SP6). Stimulation is delivered with adisperse-dense wave, 2Hz in frequency. The stimulation intensity is adjusted in accordance with the maximal level tolerated by each patient.
  Interventions: Other: transcutaneous electrical acupoint stimulation
- whole-process transcutaneous electrical acupoint stimulation(sham stimulation) (Sham Comparator): Patients are treated bilaterally at four sham acupoints of LI4, PC6, ST36 and SP6. These four pseudo-acupoints were located 1 cun ulnarlateral, and 7 cun and 9 cun proximal to Shenmen (HT7) ;and 9 cun and 12 cun proximal of Kunlun (BL60). These sham points are picked because there are no meridians or channels through these four sites. The stimulation intensity is adjusted in the lowest level felt by each patient. Other intervention details are similar to those of the experimental group.
  Interventions: Other: transcutaneous electrical acupoint stimulation sham stimulation

INTERVENTIONS:
Other: transcutaneous electrical acupoint stimulation — Electrical stimulation is performed within 24h before surgery, 30min before anesthesia induction and 3 days after surgery, each stimulation was 30min. Patients are treated bilaterally at two groups of distal acupoints: one group consisted of Hegu (LI4) and Neiguan (PC6), the other contained Zusanli (ST36) and Shanyinjiao (SP6). Stimulation is delivered with adisperse-dense wave, 2Hz in frequency. The stimulation intensity is adjusted in accordance with the maximal level tolerated by each patient.
  Arms: whole-process transcutaneous electrical acupoint stimulation
Other: transcutaneous electrical acupoint stimulation sham stimulation — Patients are treated bilaterally at four sham acupoints of LI4, PC6, ST36 and SP6. These four pseudo-acupoints were located 1 cun ulnarlateral, and 7 cun and 9 cun proximal to Shenmen (HT7) ;and 9 cun and 12 cun proximal of Kunlun (BL60). These sham points are picked because there are no meridians or channels through these four sites. The stimulation intensity is adjusted in the lowest level felt by each patient. Other intervention details are similar to those of the experimental group.
  Arms: whole-process transcutaneous electrical acupoint stimulation(sham stimulation)

SUMMARY:
The goal of this clinical trial is to evaluate the effect of whole-process transcutaneous electrical acupoint stimulation on opioid consumption after gastrointestinal laparoscopic surgery. All subjects received conventional multimodal analgesia. On this basis, the experimental group received whole-process transcutaneous electrical acupoint stimulation, while the control group received corresponding false stimulation.

DETAILED DESCRIPTION:
Conventional multimodal analgesia protocols as follows：

1. Before the end of the operation, the surgical incision was infiltrated with 0.5% ropivacaine 10 mL locally.
2. Patients were transferred to the PACU and provided with patient-controlled intravenous analgesia with sufentanil for postoperative analgesia. The analgesia devices were set to a concentration of 1ug/mL, with a lockout interval of 15 minutes, and a 3 mL bolus，without an infusion dose. The pump was withdrawn 72h after surgery.
3. Flurbiprofen: 50mg per dose intravenously twice a day for postoperative three days.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older;
* scheduled for elective laparoscopic gastrointestinal surgery；
* informed consent；
* American Society of Anesthesiologists Physical Status Grades I-III；
* body mass index (BMI) between 18.5 kg/m2 and 28 kg/m2

Exclusion Criteria:

* local skin infection, incision or scar near the study acupoints;
* nerve damage in upper or lower limbs;
* participation in other clinical trials that influence the evaluation of the results of this study;
* inability to understand the Visual Analog Scale (VAS) score or disagreeing with the use of patient controlled analgesia;
* presence of a pacemaker;
* patients with severe CNS diseases or severe mental disorders;
* operations requiring enterostomy or converts to laparotomy;
* patients who need to be transferred to the intensive care unit (ICU) for treatment after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The total sufentanil consumption postoperatively | 3 days
  measured from the recovery area until postoperative day 3

SECONDARY OUTCOMES:
The number of postoperative rescue analgesia | 7 days
  measured from the recovery area until discharge
Pain scores (VAS) | 4 days
  measured by Visual Analogue Scale( VAS ), which is a scale created in the range of 0 to 10 cm. According to the scale, 0 cm means no pain, and 10 cm means unbearable pain. On the scale, 1 to 3 cm indicates mild pain, 4 to 6 cm indicates moderate pain, and 7 to 10 cm indicates severe pain.
Pain Catastrophizing | 5 days
  measured by Pain Catastrophizing Scale（PCS）, which contains 13 items in three dimensions: rumination, magnification, and helplessness. Patients can answer on a 0-to-4 likert scale (0 = "not at all" and 4 = "all the time"). PCS scores range from 0 to 52, and the higher the score,the higher the frequency of catastrophizing cognitions.
Quality of recovery | 5 days
  measured by Quality of Recovery (QoR)-15 questionnaire, which consists of 15 questions distributed on two dimensions: "physical" and "mental" well-being. The patients report their experiences on a scale from 0 (=not at all) to 10 (=all the time), where negatively loaded questions are reversed. This gives a maximum score = 150.
The variation of C-reactive protein（CRP） | 3 days
  the values of C-reactive protein from peripheral blood
Procalcitonin（PCT） | 3 days
  the values of procalcitonin from peripheral blood
The variation of white blood cell count （WBC） | 3 days
  the values of white blood cell count from peripheral blood
Neutrophil ratio（NEUT） | 3 days
  neutrophil ratio from peripheral blood
Time to first ambulation | up to 7 days
  time to first ambulation in hours is used
Time to first flatus | up to 7 days
  time to first flatus in hours is used
Time to first defecation | 7 days
  time to first defecation in hours is used
Time to first feed | up to 7 days
  time to first feed in hours is used
The incidence rate of adverse reaction | 7 days
  adverse reaction includes PONV、abdominal distension、 diarrhea、difficult defecation ect.
Satisfaction score with pain management | 7 days
  measured by 5-point Likert scale, "1" represents very dissatisfied while "5" represents very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D.,Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China